CLINICAL TRIAL: NCT04315064
Title: Infusion of Panobinostat (MTX110) Into the Fourth Ventricle or Tumor Resection Cavity in Children and Adults with Recurrent Medulloblastoma: a Pilot Study
Brief Title: Infusion of Panobinostat (MTX110) Into the Fourth Ventricle in Children and Adults with Recurrent Medulloblastoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Midatech Pharma plc (Unknown)
Responsible Party: Principal Investigator, David Ilan Sandberg, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-19-0939
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Medulloblastoma
Keywords: medulloblastoma; Malignant Neoplasms, Brain; MTX110; panobinostat; Antineoplastic
MeSH Terms: conditions — Medulloblastoma; Brain Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with MTX110 (Experimental)
  Interventions: Drug: Treatment with MTX110

INTERVENTIONS:
Drug: Treatment with MTX110 — Patients will undergo surgery for maximum safe tumor resection with simultaneous placement of a ventricular access device (VAD) into the fourth ventricle or posterior fossa tumor resection cavity.The specific ventricular access device that will be placed is Medtronic Reference number 44102, "Medtronic CSF-Ventricular Reservoir Side Inlet, 18 mm.If a patient already has a ventricular access device in place and additional tumor resection is not required, then that patient can proceed with intraventricular chemotherapy infusions after study enrollment. If the patient has metastatic disease in the brain and/or spine without resectable tumor in the posterior fossa, then only catheter and ventricular access device placement will be performed.Enrolled patients will receive 4 infusions per week of panobinostat (MTX110; 0.25 ml of 300 μM = 26.2 μg), per infusion into the ventricular access device for 6 consecutive weeks for a total of 24 infusions.

SUMMARY:
The purpose of this study is to establish the safety of infusions of panobinostat (MTX110) into the fourth ventricle of the brain or tumor resection cavity in patients with recurrent medulloblastoma and to assess the antitumor activity of simultaneous infusions of panobinostat (MTX110) into the fourth ventricle of the brain or resection cavity in patients with recurrent medulloblastoma based upon MRI scans and lumbar cerebrospinal fluid (CSF) cytology.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Patients with histologically verified medulloblastoma with recurrence or progression involving anywhere in the brain and/or spine.
* Patient must have either measurable or evaluable tumor as assessed by MRI of the brain and total spine
* An implanted catheter in the fourth ventricle or posterior fossa tumor cavity attached to a ventricular access device or agreement to have one placed.
* A minimum of 7 days between last dose of systemic chemotherapy and/or radiation therapy and first infusion of chemotherapy into fourth ventricle
* Life expectancy of at least 12 weeks in the opinion of the principal investigator
* Lansky score of 50 or greater if ≤16 years of age or Karnofsky score of 50 or greater if > 16 years of age
* Existing neurological deficits must have been stable for a minimum of 1 week prior to study enrollment
* Patients must have recovered from the acute toxic effects of all prior anticancer chemotherapy
* Adequate bone marrow function defined by peripheral absolute neutrophil count (ANC) ≥ 500/µL, platelet count ≥ 50,000/µL (transfusion independent), and hemoglobin ≥ 9.0 gm/dL (may receive red blood cells(RBC) transfusions)
* Patient or patient's legal representative, parent(s), or guardian able to provide written informed consent.
* Patient with prolonged QT interval on screening EKG will need cardiology consultation prior to enrollment
* Patients with abnormal liver function tests (ALT, Aspartate Aminotransferase(AST),or total bilirubin) will need gastroenterology consultation prior to enrollment

Exclusion Criteria:

* Enrolled in another treatment protocol
* Has received another investigational or chemotherapy agent or radiation therapy within 7 days prior to intraventricular chemotherapy infusions
* Evidence of untreated infection
* Pregnant or lactating women

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with grade 3 through grade 5 new neurological adverse events that are related to study drug | 4 months post intervention
  Anew neurological deficit will be defined as new cranial neuropathy, change in level of consciousness, motor weakness, gait change or cerebellar finding (ataxia, dysmetria, dysdiadochokinesis) and will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0

SECONDARY OUTCOMES:
Change in disease progression as measured by an MRI | prior to first infusion; after last infusion (last infusion is about 6 weeks after the first infusion)
  Change in disease progression as measured by an MRI
Change in disease progression as measured by lumbar CSF cytology | prior to first infusion; after last infusion (last infusion is about 6 weeks after the first infusion)
  Change in disease progression as measured by lumbar CSF cytology

CONTACTS AND LOCATIONS:
Overall Officials: David IIan Sandberg, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No